CLINICAL TRIAL: NCT06590610
Title: Evaluation of the Independent Temporary Effects of Intelect® RPW2 (Radial Pressure Wave) and Cefar TENS (NMES) Treatments on the Local Circuclation of Healthy Volunteers
Brief Title: Post-Market Clinical Follow-up HVS on Increased Circulation, RPW2 and Cefar TENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DJO UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENOVIS-S-INP-0007
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: NMES; RPW2; CEFAR TENS; healthy volunteers; haemodynamic changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- electrotherapy (Experimental): All the selected 20 healthy subjects will undergo the radial pressure waves treatment on one leg at the Gastrocnemius, left or right leg as per randomization. Afterwards each patient will undergo NMES electrostimulation treatment on the opposite leg at the Gastrocnemius.
  Interventions: Device: Radial pressure wave (RPW) - Intelect RPW2 Chattanooga

INTERVENTIONS:
Device: Radial pressure wave (RPW) - Intelect RPW2 Chattanooga — RPW treatment on one leg at the Gastrocnemius and NMES electrostimulation on the opposite leg. RPW or NMES treatment on each leg will be randomized prior to application with each device having an equal chance of being placed on the either leg (dominant and non-dominant).
  Other Names: NMES electrostimulation - CEFAR TENS Chattanooga

SUMMARY:
The study is a prospective, single-center, open-label, post-market investigational study on healthy volunteers conducted in the United Kingdom.

Sponsor is conducting this prospective study to collect PMCF data on the safety and performance of Intelect RPW2 and CEFAR TENS devices in accordance with Medical Device Regulation (EU) 2017/745 (MDR) Article 61 and Part B of Annex XIV.

The aim of this study is to measure the hemodynamic changes in the lower limb consequent to the use of CEFAR TENS via neuromuscular electrical stimulation (NMES) and to the use of Intelect® RPW2 via radial pressure waves (RPW).

The hypothesis of this study is that the application of both medical devices, CEFAR TENS or Intelect® RPW2 to the calf muscles will increase venous return, as a local and temporary effect of the treatment.

The hemodynamic measurements will be recorded with a Duplex ultrasound at baseline before the treatment as steady state condition, during the treatment session at several timepoints and after each treatment's end.

DETAILED DESCRIPTION:
The selected 20 healthy subjects will undergo one treatment per device for both electrostimulation and radial pressure wave therapy on both the right and left Gastrocnemius, device placement on each leg will be randomized prior to application with each device having an equal chance of being placed on the either leg (dominant and non-dominant). Each subject will receive treatment via the Intelect® RPW2 device to either the right or left leg and afterwards the subject will receive treatment via the CEFAR TENS device to the opposite leg as per the randomization table.

The capability of the radial pressure waves therapy (Intelect® RPW2) and NMES (CEFAR TENS) to improve local and temporarily hemodynamics on the treated limb will be investigated.

The subject will firstly receive RPW treatment and secondly receive NMES treatment this will be consistent for all subjects, as an arbitrary decision to be consistent throughout the whole study with the treatment's application.

Subjects will be positioned in the prone decubitus position for a minimum of 3 minutes or until the steady state condition is reached; automated blood pressure cuff will be used to record blood pressure and pulse from upper arm. Following the rest period the measurement by means of a Duplex Ultrasound will be performed: Peak venous velocity, Ejected volume, Time averaged Mean venous velocity, and Volume flow will be recorded in the leg to be treated with RPW. Subjects will remain in this position for the duration of the treatment (corresponding to 2 minutes and 30 seconds by RPW and 10 minutes for NMES), the study staff will apply the Intelect® RPW2 device to either the right or left leg according to the randomization plan. During the RPW treatment the hemodynamic parameters in the subject leg will be measured at 30 seconds, 1 minute, 1 minute and 30 seconds, 2 minutes and 2 minutes and 30 seconds after RPW treatment is started and at 1, 2, 5 and 10 minutes after RPW treatment end. Arterial blood pressure and heart rate measurement will be recorded after RPW treatment end from upper arm.

Then the study staff will apply the CEFAR TENS device to the opposite leg. During the NMES treatment the hemodynamic parameters in the subject leg will be measured at 30 seconds, 1, 2 ,5, 8 and 10 minutes after NMES treatment is started and at 1, 2, 5 and 10 minutes after treatments end. Blood pressure and pulse will be recorded after NMES treatment end from upper arm.

The treatment with Intelect® RPW2 and CEFAR TENS devices will be performed by the study staff after training on the devices use.

A Vascular Technologist will perform the hemodynamic measurements by Duplex Ultrasound device.

A virtual follow up visit will be scheduled one week following treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, both male and female, ≥ 18 years of age at the time of consent.
2. Subject is available to attend all study appointments for the study duration
3. Any Subject who has reviewed the IEC-approved consent form, has been properly consented per the protocol and has documented their consent to participate in the study by signing the Ethics-approved consent form.

Exclusion Criteria:

1. Subjects with any cognitive impairment who prevent to understand the information provided and freely and autonomously provide and sign informed consent to participate in the study.
2. Subject is pregnant or has plans of becoming pregnant for the duration of the study.
3. Presence of cancerous tumours/Neoplastic tissue/lesions in treatment area (back lower limb of both legs)
4. Subject possesses a prosthetic lower limb
5. Diagnosed with diabetes
6. Cortisone therapy ongoing or within the last 6 months before treatment
7. Diagnosed Haemophilia, Thrombosis, Deep vein thrombosis, phlebitis, varices, risk of haemorrhage, occlusive vascular disease or other coagulation disorders
8. Treatment with anticoagulant pharmaceuticals
9. Reduced sensitivity over the proposed area of treatment (back lower limb of both legs)
10. Suspected or diagnosed cardiopathy
11. Any history of cardiovascular disease e.g., cardiac arrhythmia and angina pectoris, arterial disease, circulatory insufficiency.
12. Implanted electronic devices e.g., cardiac stimulator, implanted defibrillator or other implanted electronic/electrical device
13. Hypertension (> stage 2), ischemic heart disease and cerebrovascular diseases
14. Peripheral vascular disease or serious arterial or venous circulation problems in any of the lower limbs.
15. Systemic or local infection.
16. Open wounds, rashes, swollen, red, infected, inflamed areas or skin eruptions at the site of treatment (back lower limb of both legs).
17. Diagnosis of Epilepsy or has had any previous Epileptic episodes.
18. Proven allergy to the study devices materials or electrodes.
19. Recent surgery or metal implant present at the site of treatment (back lower limb of both legs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
PV - Peak venous velocity (cm/s) will be assessed by Duplex Ultrasound (Philips EPIQ 7) | PV assessment will be on the same day of the RPW treatment: before, during, and at treatment's end on one leg. PV assessment will be on the same day of the NMES treatment: before, during, and at treatment's end on the opposite leg.
  PV is here defined as primary endpoint to verify the hypothesis of hemodynamic changes and blood flow improvements due to the applied treatments with the devices under investigation within this study.
  The effects of the application of CEFAR TENS and Intelect® RPW2 on the calf muscles on local peak venous velocity will be compared to steady state values. The comparison between the hemodynamic measurements collected during and following each treatment has been performed and the pre-treatment steady state values will provide evidence of the hemodynamic changes hypothesized

SECONDARY OUTCOMES:
EV - Ejected volume (ml) will be assessed by Duplex Ultrasound (Philips EPIQ 7) | EV assessment will be on the same day of the RPW treatment: before, during, and at treatment's end on one leg. EV assessment will be on the same day of the NMES treatment: before, during, and at treatment's end on the opposite leg
  This secondary endpoint has been identified as parameter commonly evaluated in the scientific literature on similar studies to evaluate the beneficial effect of NMES treatment on blood circulation.
Time averaged Mean venous velocity (cm/s) will be assessed by Duplex Ultrasound (Philips EPIQ 7) | Velocity assessment will be on the same day of the RPW treatment: before, during, and at treatment's end on one leg.Velocity assessment will be on the same day of the NMES treatment: before, during, and at treatment's end on the opposite leg
  This secondary endpoint has been identified as parameter commonly evaluated in the scientific literature on similar studies to evaluate the beneficial effect of NMES treatment on blood circulation.
Volume flow (VF) in mL/min will be assessed by Duplex Ultrasound (Philips EPIQ 7) | Volume flow assessment will be on the same day of the RPW treatment: before, during, and at treatment's end on one leg.Volume flow assessment will be on the same day of the NMES treatment: before, during, and at treatment's end on the opposite leg
  This secondary endpoint has been identified as parameter commonly evaluated in the scientific literature on similar studies to evaluate the beneficial effect of NMES treatment on blood circulation.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Whiteley, MD, Surgeon, Principal Investigator — The Whiteley Clinic
Locations (1):
- The Whiteley Clinic, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No